CLINICAL TRIAL: NCT06429592
Title: The Effect of the Empowerment Program Constructed According to Neuman's Systems Model on Stress and Satisfaction Levels of Mothers With Children in the Intensive Care Unit and Effective Decision Making
Brief Title: Stress and Satisfaction Levels of Mothers According to Neuman's Systems Model on Stress and Satisfaction Levels of Mothers With Children in the Intensive Care Unit and Effective Decision Making
Status: Not yet recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gulsah Ogul, Principal Investigator, TC Erciyes University
Other Study IDs: gulsahogulerciyes4023640013
Record Dates: First submitted 2024-05-20; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Nurse-Patient Relations
Keywords: Mother; Pediatric intensive care; Effective decision making; Satisfaction; Stres
MeSH Terms: conditions — Personal Satisfaction | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Data collection tools for mothers in the experimental group after acceptance of admission to the intensive care unit [Descriptive Characteristics Form, Parental Stress Scale: (Pediatric Intensive Care Unit), Empowerment of Parents in The Intensive Care (EMPATHIC-30) (Empowerment of Parents in Intensive Care Scale), Decision Data will be collected using the Conflict in Making and Decision Making Confident Scale (KVÇS and KEOÖ). The prepared strengthening program will be applied for a total of 5 days starting from the first day of hospitalization. While the mothers are being treated, no other treatment will be done in the unit.
  Different time slots will be scheduled for each experiment. After the 5th day of the application was completed, data collection tools were used.
  Interventions: Other: education
- control group: Data collection tools from mothers in the control group after admission to the intensive care unit [Descriptive Characteristics Form, Parental Stress Scale: (Pediatric Intensive Care Unit), Empowerment of Parents in The Intensive Care (EMPATHIC-30) (Empowerment of Parents in Intensive Care Scale), Decision Data will be collected using the Conflict in Making and Decision Making Confident Scale (KVÇS and KEOÖ). The routine operation of the intensive care unit will continue and data will be collected again after 5 days of hospitalization.
  Interventions: Other: education

INTERVENTIONS:
Other: education — nursing care practice

SUMMARY:
Research; It will be carried out to examine the effect of the empowerment program structured according to the Neuman systems model on the stress and satisfaction levels and effective decision-making of mothers whose children are in the intensive care unit.

DETAILED DESCRIPTION:
For pediatric nurses, supporting families, especially mothers, who take a primary role in care, increasing their ability to cope with the stress they experience, helping them access the information and resources they need, and supporting family functionality are vital parts of nursing care.

In order to strengthen the family, the relationship between the nurse and the family must be based on respect and trust. In the nurse's communication with the family; The family should discuss the expectations of the family, discuss their views, and care about how much the family wants to be involved in care and what they want to do. Communication provided through these foundations helps to establish a trusting relationship between the family and the nurse and to determine boundaries with the parents. In this way, role confusion between the nurse and parent can be prevented and bidirectional satisfaction can be achieved.

Another issue required to strengthen the family is to establish a close physical and emotional bond between the nurse and the family. This bond is related to the family feeling close enough to the nurse to open up to them not only in the presence of the problem, but also outside the problems. Thus, the family's trust in the nurse increases, removing the nurse from the position of healthcare personnel only caring for the child. Thanks to this special bond the nurse establishes with the family, it makes it easier for family members to express themselves and can even help them discover their weaknesses that they are not aware of. In addition, the nurse evaluates the family's coping methods, helps reveal their strengths, and can ensure more effective planning of care. Studies have shown that as a result of the empowerment programs applied by nurses to families, parents' depression and stress levels decrease, family function, self-efficacy, autonomy, problem-solving skills and family members' support for each other increases.

In order to strengthen the family, it is of great importance to reduce the effects of internal and external stressors, holistic approach, increase the patient's perceptions and motivation, interact with the environment, reach, protect and maintain optimal health. In line with this purpose, the conceptual framework of nursing theories and models forms the basis and directs nursing education, management, practice and nursing research. These components are also included in the philosophical basis of the Neuman Systems Model. Neuman Systems Model is a model that focuses on human needs and emphasizes human uniqueness. It focuses on the multidimensional evaluation of the individual from a holistic perspective in achieving optimal health/well-being. However, accepting that the human being is a biopsychosocial being, it attaches importance to environmental stress and the health of the patient system that reacts to this stress. In Neuman's Systems Model, it is stated that when an individual is exposed to various stressors, his defense system is affected and the individual needs help to protect his basic structure.

It is thought that nursing care structured in line with the Neuman Systems Model facilitates family and child-centered care practice. This study will be conducted to examine the effect of the empowerment program structured according to the Neuman systems model on the stress and satisfaction levels and effective decision-making of mothers whose children are in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Research Inclusion Criteria;

  1. Communicable,
  2. Mothers whose children are admitted to the intensive care unit,
  3. Mother must be over 18 years old
  4. The child has a biological mother
  5. Mothers who agreed to participate in the study and signed written consent forms,
  6. The child's intensive care stay must be at least 5 days.

Exclusion Criteria:

* Criteria for Exclusion from the Study

  1. Wanting to leave the study,
  2. The child must have left the intensive care unit less than 5 days ago,
  3. The mother is under 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers who want to voluntarily participate in the research
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-17 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Mothers' stress levels and satisfaction levels will be evaluated. | 3 months
  For mothers in the experimental group, data will be collected with data collection tools after acceptance of admission to the intensive care unit. The prepared strengthening program will be applied for a total of 5 days starting from the first day of hospitalization. While the treatments are being carried out to the mothers, no other treatments will be performed in the unit.
  Different time slots will be scheduled for each experiment. After the 5th day of the application is completed, data will be collected with data collection tools and mothers' stress levels and satisfaction levels will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: oznur basdas, professor, Study Director — erciyes universitesi